CLINICAL TRIAL: NCT07146880
Title: Empagliflozin as a Potential Therapeutic Solution for Patients With Brugada Syndrome
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202506158MINB
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Brugada Syndrome (BrS)
Keywords: Brugada Syndrome (BrS); Sodium-glucose cotransporter 2 inhibitors (SGLT-2i); Empaflifozin
MeSH Terms: conditions — Brugada Syndrome | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Empagliflozin (Experimental)
  Interventions: Drug: Empagliflozin (EMPA)

INTERVENTIONS:
Drug: Empagliflozin (EMPA) — Participants will take Empagliflozin once daily, starting at 10 mg. The dose will be increased to 25 mg at monthly follow-ups if participants are non-responders based on ECG ST-segment morphology. The total treatment period is three months.

SUMMARY:
The goal of this clinical trial is to learn if Empagliflozin works to treat Brugada syndrome patients by affecting their electrocardiographic (ECG) patterns, and to evaluate its safety.

The main questions it aims to answer are:

* Does Empagliflozin improve specific electrocardiogram (ECG) patterns in Brugada syndrome patients, specifically by observing the change in J-point elevation recorded in V1 and V2 leads at the 4th, 3rd, and 2nd intercostal spaces (ICSs)? A responder is defined as a decrease in J-point elevation of ≥1 mm.
* What adverse events do participants experience when taking Empagliflozin, including hypotension, acute renal failure, hepatic injury, ketoacidosis, hypoglycemic events, urinary tract infections, genital infections, bone fractures, and events leading to lower limb amputation?

Researchers will compare each participant's ECG changes before and after three months of Empagliflozin treatment to assess its efficacy

Participants will:

* Take Empagliflozin once daily, starting at 10 mg. The dose will be increased to 25 mg at monthly follow-ups if participants are non-responders based on ECG ST-segment morphology. The total treatment period is three months.
* Visit the outpatient clinic monthly for three months of treatment to monitor efficacy and safety. The overall trial period, including screening, treatment, and follow-up, comprises five scheduled visits.
* Undergo a series of check-ups and tests, including:

  * 12-lead electrocardiography (ECG) recordings.
  * Monitoring and documentation of adverse events.
  * Blood and urine tests, such as complete blood count (CBC), liver function tests (AST/ALT), renal function tests (BUN/creatinine), electrolytes (sodium/potassium/calcium/magnesium/albumin), urinalysis, fasting glucose, HbA1c, and ketone measurements.

DETAILED DESCRIPTION:
Inclusion Criteria

1. Patients diagnosed with Brugada syndrome and aged 18-99 years with spontaneous type 1 ECG, normal structural heart and patent coronary artery
2. Obtain written informed consent for participation in the clinical trial

Exclusion Criteria

1. Individuals with type 1 ECG pattern only observed with fever-induced or drug-induced were excluded from this exploratory study.
2. Current or prior use of an SGLT2 inhibitor within 12 weeks before screening or randomization
3. Known allergy or hypersensitivity to any SGLT2 inhibitor
4. History of ketoacidosis
5. Symptomatic hypotension or systolic blood pressure <90 mmHg or >180 mmHg
6. Heart failure
7. Acute myocardial infarction
8. ALT or AST >3× ULN at screening
9. Impaired renal function (eGFR <20 mL/min/1.73 m² [MDRD]), requiring dialysis, or functioning kidney transplant at screening
10. Pregnancy, nursing, or planning pregnancy during the trial
11. Enrollment in another investigational drug or device study or completion of such a study within the last 30 days
12. Known poor adherence to clinic visits or prescribed medications
13. Medical conditions that may limit trial participation, including severe respiratory disease, history of cancer with metastasis in the past four years (excluding non-melanoma skin cancer), or recent alcohol/substance misuse

Trial protocol The initial dose will start at 10 mg empagliflozin once a day, with monthly follow-ups for dose titration based on ECG ST-segment morphology done in lead V1, V2 at 4th, 3rd and 2nd intercostal spaces (ICSs). Responder is defined as any one of lead with a decrease in J-point elevation ≥1 mm from baseline. Responders will continue receiving 10 mg empagliflozin once a day, while non-responders will have their dose increased to 25 mg once a day.

This study followed a structured clinical trial protocol, including Screening, Treatment, and Follow-up periods. Participants underwent assessments at five scheduled visits corresponding to weeks -4 (screening), 4, 8, 12 (treatment phase), and 16 (follow-up). Peripheral blood mononuclear cell，(PBMC) will be collected and send to Stanford lab for Induced pluripotent stem cell (iPCS) once patient is enrolled in this study. Key evaluations included body weight (BW), automated office blood pressure (AOBP), and 12-lead electrocardiography (ECG). Safety monitoring encompassed adverse event documentation and laboratory tests with 15ml blood sample, including complete blood count (CBC), liver function tests (AST/ALT), renal function tests (BUN/creatinine), urinalysis, glucose AC, HbA1c, and ketone measurements. These assessments were conducted at predefined time points to ensure comprehensive monitoring of treatment effects and safety throughout the study duration.

Endpoints

Efficacy Endpoint Maximal change of type 1 Brugada ECG pattern recording with lead V1 and V2 in 4th, 3rd, and 2nd ICSs. Change of type 1 Brugada ECG pattern was defined as maximal J point elevation minus baseline J point elevation in the same leads. The responder is defined as decreased ≥ 1mm of J point in any one of above 6 leads.

Safety Endpoint Adverse event (AE) will be monitored as trail protocol. Adverse event including hypotension, symptomatic hypotension, acute renal failure, hepatic injury, ketoacidosis, hypoglycemic events, urinary tract infections, genital infections, bone fractures, events leading to lower limb amputation.

A serious adverse event (SAE) is any adverse event that results in death, is life-threatening, necessitates hospitalization or prolongation of existing hospitalization, causes significant disability or incapacity, leads to congenital anomalies or birth defects, or is deemed medically significant, potentially requiring intervention to prevent serious outcomes.

In accordance with the study protocol, the hospital will provide professional medical care and consultation in the event of adverse reactions or harm resulting from the clinical trial. Any adverse events will be reported to the Institutional Review Board (IRB) as required, with continuous monitoring of other participants' responses. All tests conducted are routine hospital examinations and pose no psychological harm to participants. Participant rights and protections will be upheld in accordance with the informed consent agreement.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Brugada syndrome and aged 18-99 years with spontaneous type 1 ECG, normal structural heart and patent coronary artery
2. Obtain written informed consent for participation in the clinical trial

Exclusion Criteria:

1. Individuals with type 1 ECG pattern only observed with fever-induced or drug-induced were excluded from this exploratory study.
2. Current or prior use of an SGLT2 inhibitor within 12 weeks before screening or randomization
3. Known allergy or hypersensitivity to any SGLT2 inhibitor
4. History of ketoacidosis
5. Symptomatic hypotension or systolic blood pressure <90 mmHg or >180 mmHg
6. Heart failure
7. Acute myocardial infarction
8. ALT or AST >3× ULN at screening
9. Impaired renal function (eGFR <20 mL/min/1.73 m² [MDRD]), requiring dialysis, or functioning kidney transplant at screening
10. Pregnancy, nursing, or planning pregnancy during the trial
11. Enrollment in another investigational drug or device study or completion of such a study within the last 30 days
12. Known poor adherence to clinic visits or prescribed medications
13. Medical conditions that may limit trial participation, including severe respiratory disease, history of cancer with metastasis in the past four years (excluding non-melanoma skin cancer), or recent alcohol/substance misuse

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-08-21 (Estimated); Study Completion 2027-09-21 (Estimated)

PRIMARY OUTCOMES:
Maximal change of type 1 Brugada pattern (defined as maximal J point deviation minus baseline J point hight) recording with 12-lead electrocardiogram within lead V1 and V2 in 4th, 3rd, and 2nd ICSs | From enrollment to the end of treatment at 8 weeks
  Maximal Change of type 1 Brugada pattern (Coved ST segment elevation >2mm in >1 of V1-V3 followed by a negative T wave.) is defined as maximal J point deviation minus baseline J point elevation in the same leads. The responder is defined as decreased ≥ 1mm of J point in any one of above 6 leads.

OTHER OUTCOMES:
Incidence of Treatment-Related Adverse Events (Safety and Tolerability) | From enrollment to the end of tial at 12 weeks
  Adverse event (AE) will be monitored as trail protocol. Adverse event including hypotension, symptomatic hypotension, acute renal failure, hepatic injury, ketoacidosis, hypoglycemic events, urinary tract infections, genital infections, bone fractures, events leading to lower limb amputation.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Wu, MD, Phd, Principal Investigator — Stanford University; JYH-MING JIMMY JUANG, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No